CLINICAL TRIAL: NCT01642121
Title: Observational - Rapid Identification of Leukemia Stem Cells Associated With AML1-ETO and Inv(16) Through Characterization of Oncogene-Induced Changes in Cell-Surface Antigen Profiles on Hematopoietic Stem Cells
Brief Title: Studying Biomarkers in Samples From Younger Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML12B10; NCI-2012-01983 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Acute Monoblastic Leukemia (M5a); Childhood Acute Monocytic Leukemia (M5b); Childhood Acute Myeloblastic Leukemia Without Maturation (M1); Childhood Acute Myeloid Leukemia/Other Myeloid Malignancies; Childhood Acute Myelomonocytic Leukemia (M4)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Samples and controls are sorted and re-sorted for CD34, CD38, and CD55 subsets by single-cell PCR analysis, flow cytometry, and reverse-transcriptase PCR. Sorted cell subsets are then transplanted into NSG mice. Beginning 6 weeks after transplantation, peripheral blood samples are collected and analyzed for human lymphoid- and myeloid-lineage cells by FACS.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This laboratory study is looking into biomarkers in samples from younger patients with acute myeloid leukemia. Studying samples of bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer

DETAILED DESCRIPTION:
Study Subtype: Observational Observational Study Model: Case-control Time Perspective: Retrospective Biospecimen Retention: Samples With DNA Biospecimen Description: Cryopreserved bone marrow samples Study Population Description: Patient samples with the AML1-ETO translocation and cytologically normal AML samples for controls Sampling Method: Non-Probability Sample

OBJECTIVES:

I. To address whether the mutation-specific cell-surface markers observed in murine system will allow the prospective isolation of leukemia stem cells (LSC) from human bone marrow samples that have the same cytogenetic abnormalities.

II. To compare the incidence of leukemia in NSG mice that have received CD34+CD38 marker+ cells to NSG mice that receive what are hypothesized to be normal cells (CD34+CD38 marker-subset) from the same patient.

OUTLINE:

Samples and controls are sorted and re-sorted for CD34, CD38, and CD55 subsets by single-cell polymerase chain reaction (PCR) analysis, flow cytometry, and reverse-transcriptase PCR. Sorted cell subsets are then transplanted into NSG mice. Beginning 6 weeks after transplantation, peripheral blood samples are collected and analyzed for human lymphoid- and myeloid-lineage cells by fluorescence-activated cell sorting (FACS).

ELIGIBILITY:
Inclusion Criteria:

* Frozen bone marrow aspirates obtained from childhood acute myeloid leukemia (AML) patients possessing defined cytogenetic mutations; AML1-ETO or inv(16)
* Samples of cytogenetically normal AML cases obtained from the University of Alabama at Birmingham (UAB) as controls

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: childhood acute myeloid leukemia (AML) patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Expression of the CD55 marker on CD34+CD38- cells | Up to 6 months
Presence of the AML1-ETO translocation | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Heidemann, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States